CLINICAL TRIAL: NCT04176952
Title: PRIMUS002: An Umbrella Phase II Study Examining Two Neo-adjuvant Regimens (FOLFOX-A and AG) in Resectable and Borderline Resectable Pancreatic Ductal AdenoCarcinoma (PDAC), Focusing on Biomarker and Liquid Biopsy Development
Brief Title: PRIMUS002: Looking at 2 Neo-adjuvant Treatment Regimens for Resectable and Borderline Resectable Pancreatic Cancer
Acronym: PRIMUS002
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to funding being withdrawn
Sponsor: Judith Dixon-Hughes (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other); University of Glasgow (Other)
Responsible Party: Sponsor-Investigator, Judith Dixon-Hughes, Project Manager, University of Glasgow
Organization: University of Glasgow (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRIMUS0022016
Record Dates: First submitted 2019-10-28; First posted 2019-11-26 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Neoplasms Pancreatic
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients are registered to receive either FOLFOX-A or AG depending on their age and performance status
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOLFOX-A (Experimental): FOLFOX A arm (14-day cycle)
  * nab-paclitaxel: 150mg/m2 IV over 30 minutes, day 1 (administered first).
  * Oxaliplatin: 85mg/m2, IV over 2 hours, day 1.
  * Folinic acid: 350mg flat dose, IV over 2 hours, day 1.
  * Fluorouracil infusion:1200mg/m2/day, as a continuous IV infusion over 2 days, day 1 and day 2 (for a total dose of 2400mg/m2 over 46 hours or 48 hours as per local practice.)
  Patients will also receive daily G-CSF as primary prophylaxis against neutropenic events for all cycles. This should be given as per local policy for chemotherapy regimens given every 14 days e.g. it may be started on day 4 for 7 days (preparation and dose should be given as per local policy).
  Interventions: Drug: FOLFOX-A
- Abraxane and Gemcitabine (Active Comparator): Nab-Paclitaxel + Gemcitabine (AG) arm (28-day cycle)
  * nab-paclitaxel: 125mg/m2 IV over 30 minutes on days 1, 8 and 15 (administered first).
  * Gemcitabine 1000mg/m2 IV over 30 minutes on days 1, 8 and 15 (immediately following nab-paclitaxel).
  Interventions: Drug: AG

INTERVENTIONS:
Drug: FOLFOX-A — * nab-paclitaxel: 150mg/m2 IV over 30 minutes, day 1 (administered first).
  * Oxaliplatin: 85mg/m2, IV over 2 hours, day 1.
  * Folinic acid: 350mg flat dose, IV over 2 hours, day 1.
  * Fluorouracil infusion:1200mg/m2/day, as a continuous IV infusion over 2 days, day 1 and day 2 (for a total dose of 2400mg/m2 over 46 hours or 48 hours as per local practice.)
  Arms: FOLFOX-A
Drug: AG — * nab-paclitaxel: 125mg/m2 IV over 30 minutes on days 1, 8 and 15 (administered first).
  * Gemcitabine 1000mg/m2 IV over 30 minutes on days 1, 8 and 15 (immediately following nab-paclitaxel).
  Arms: Abraxane and Gemcitabine

SUMMARY:
PRIMUS 002 is looking at 2 different chemotherapy regimens in the neo-adjuvant setting for pancreatic cancer. Each treatment will be given for 3 months prior to surgery

DETAILED DESCRIPTION:
This is an integrated, open label, non-randomised, phase II trial of 2 neo-adjuvant regimens (FOLFOX-A and AG) assessing efficacy and toxicity with integrated translational work. The study is powered on testing a proposed DNA damage response deficient biomarker for responsiveness in patients treated with FOLFOX-A; patients being treated with AG are recruited concurrently. The study has a prospective safety assessment of neo-adjuvant chemotherapy and neo-adjuvant chemotherapy followed by chemoradiotherapy consisting of conventional radiotherapy with concomitant capecitabine. This safety assessment will include all patients (FOLFOX-A and AG)

ELIGIBILITY:
Inclusion Criteria:

1. Patient has been enrolled in the Precision-Panc Master Protocol and their tissue has been deemed suitable for Next Generation Sequencing analysis (a Precision-Panc Master Protocol identifier will be required at the time of study enrolment)
2. Signed informed consent given for PRIMUS 002 study
3. Age ≥ 16 years
4. Resectable or borderline resectable pancreatic cancer as defined by National Comprehensive Cancer Network criteria following discussion at the Multi Disciplinary Team
5. Measurable Disease as per RECIST 1.1
6. Histological or cytologically proven pancreatic ductal adenocarcinoma (including variants)
7. Able to undergo biliary drainage using a covered or partially covered self-expanding metal stent if jaundiced
8. Eastern Cooperative Oncology Group performance status 0 and 1
9. Adequate liver/bone marrow function as defined by:

   1. Neutrophils (ANC) ≥ 1.5 x 109/l
   2. Platelets ≥ 100 x 109/l
   3. Haemoglobin ≥ 9.0g/dL
   4. White Blood Cells (WBC) ≥ 3 x 109/l
   5. Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) unless bilirubin rise is due to Gilbert's syndrome
   6. Aspartate transaminase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN (or <5 x ULN in the presence of liver metastases)
   7. Estimated creatinine clearance ≥ 60 mL/min (as calculated by Cockcroft and Gault or Wright formula or measured by EDTA clearance)
10. Negative serum Human Chorionic Gonadotropin (HCG) test for females with child bearing potential. Postmenopausal women must have been amenorrhoeic for at least 12 months to be considered of non-childbearing potential
11. Woman of child bearing potential, and men with female partners of child bearing potential, must agree to use adequate contraceptive measures (see section 7.1.11.1) for the duration of the study and for up to 6 months after the completion of study treatment.
12. Able to comply with protocol requirements and deemed fit for surgical resection, chemotherapy and CRT

Exclusion Criteria:

1. Distant metastatic disease
2. History of previous or concurrent malignancy diagnosis (except curatively treated basal cell carcinoma of skin or carcinoma in situ of cervix) in the last 3 years
3. Prior chemotherapy or CRT for pancreatic cancer
4. Known hypersensitivity for any component of any study drug
5. Active infection including Herpes Zoster and chickenpox
6. Uncontrolled congestive heart failure (CHF), or history of myocardial ischemia (MI), unstable angina, stroke, or transient ischemia within previous 6 months.
7. Serious medical or psychological condition precluding neo-adjuvant treatment and surgical resection
8. New York Heart Association Classification Grade III or IV
9. Liver cirrhosis (except for Child-Pugh A)
10. Major surgery within 28 days prior to trial entry
11. Any patients receiving treatment with brivudin, sorivudin and analogues or patients who have not stopped these drugs at least 4 weeks prior to the start of study treatment
12. Any patient with severe diarrhoea (defined as ≥grade 3 diarrhoea despite maximum supportive measures and exclusion of underlying infection)
13. Patients with known malabsorption
14. Patients with known or suspected dihydropyrimidine dehydrogenase (DPD) deficiency
15. Grade ≥ 2 peripheral neuropathy
16. Administration of any investigational drug within 28 days or 5 half-lives, whichever is longer, prior to receiving the first dose of trial treatment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Time to progression post FOLFOX-A induction treatment | CT scans will take place at baseline, pre chemoradiotherapy and pre surgery, over approximately 6 months
  date of progression after FOLFOX-A neo-adjuvant chemotherapy as assessed by RECIST 1.1

SECONDARY OUTCOMES:
Proving liquid biopsies can be used to define patient subgroups | From date of registration to date of surgery. On average 4 months after registration
  a liquid biopsy will be taken and analysed using circulating tumour DNA at different timepoints to see if these can be used to define patient subgroups
Response post neo-adjuvant chemotherapy | CT scan will be performed at baseline and then post neo-adjuvant chemotherapy (approximately 3 months later)
  CT scans will be reported to RECIST 1.1 and best response will be evaluated
College of American Pathologists tumour regression grade | Post surgery which will be approximately 4 months post registration
  CAP tumour regression grade (grade 0-3 with 0 being no viable residual tumour and 3 being poor to no response) will be assessed post surgery
R0 rate post surgery | Post surgery which will be approximately 4 months post registration
  R0 rate will be assessed post surgery
Overall survival | From date of registration until date of death assessed for up to 5 years post registration
  Overall survival will be assessed in all patients
Disease free survival | from date of registration until date of disease recurrence assessed for at least 24 months post registration
  Disease free survival will be assessed at every follow up visit
Safety and tolerability of study drugs: NCI CTCAE 4.03 | Assessed at every clinic visit during treatment, for approximately 3 months post registration
  Safety and tolerability will be assessed as per NCI CTCAE 4.03
Safety and tolerability of chemoradiotherapy: NCI CTCAE 4.03 | Assessed at every chemoradiotherapy visit and pre-surgery (once Chemoradiotherapy added). Chemoradiotherapy will take place 5 days a week for three weeks
  Safety and tolerability of chemoradiotherapy will be assessed as per NCI CTCAE 4.03
Surgical complication rate | Assessed post surgery, approximately 4 months post registration
  Rate of surgical complication as assessed by NCI CTCAE 4.03
Neurotoxicity | Neurotoxicity will be assessed from registration until study is completed at various timepoints until patient death. Each patient will be followed up for at least 24 months post registration
  Assessed by GOG NTX4 (4 questions graded from 0 (not at all) to 4 (very much). quality of life will be assessed using the GOG NTX4 tool at the following timepoints: Baseline, month 1, month 2, month 3, pre chemoradiotherapy, between fraction 11 and 15 of chemoradiotherapy, pre surgery, at every follow-up visit (6, 9, 12 months post registration then every 6 months)
Quality of life assessed by EORTC QLQ-C30 | Quality of life will be assessed from registration until study is completed at various timepoints until patient death. Each patient will be followed up for at least 24 months post registration
  quality of life will be assessed using the EORTC QLQ C30 tool at the following timepoints: Baseline, month 1, month 2, month 3, pre chemoradiotherapy, between fraction 11 and 15 of chemoradiotherapy, pre surgery, at every follow-up visit (6, 9, 12 months post registration then every 6 months for a minimum of 24 months). The Quality of life tool is comprised of 28 questions that the patient answers either 1-4 (1 = not at all, 4 = Very much) and 2 questions that are on al scale of 1 - 7 where 1 = very poor and 7 = excellent
Quality of life assessed by EORTC QLQ-PAN26 | Quality of life will be assessed from registration until study is completed at various timepoints until patient death. Each patient will be followed up for at least 24 months post registration
  quality of life will be assessed using the EORTC QLQ-PAN26 tool at the following timepoints: Baseline, month 1, month 2, month 3, pre chemoradiotherapy, between fraction 11 and 15 of chemoradiotherapy, pre surgery, at every follow-up visit (6, 9, 12 months post registration then every 6 months for a minimum of 24 months). The Quality of life tool is comprised of 26 questions that the patient answers either 1-4 (1 = not at all, 4 = Very much)
Health Economics | Health economics will be assessed from registration until study is completed at various timepoints until patient death. Each patient will be followed up for at least 24 months post registration
  Health economics defined as number of visits to hospital per patient, both as an inpatient and as an outpatient will be assessed at the following timepoints: Baseline, month 1, month 2, month 3, pre chemoradiotherapy, between fraction 11 and 15 of chemoradiotherapy, pre surgery, at every follow-up visit (6, 9, 12 months post registration then every 6 months for a minimum of 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Grose, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (3):
- United Kingdom (3):
  - Western General, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Free Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Clinical data will be made available on request once clinical study report has been written and primary publication accepted by peer reviewed journal
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Once clinical study report has been written and primary publication accepted by peer reviewed journal
Access Criteria: On request to trial management group

REFERENCES:
- [Derived] Saha A, Wadsley J, Sirohi B, Goody R, Anthony A, Perumal K, Ulahanan D, Collinson F. Can Concurrent Chemoradiotherapy Add Meaningful Benefit in Addition to Induction Chemotherapy in the Management of Borderline Resectable and Locally Advanced Pancreatic Cancer?: A Systematic Review. Pancreas. 2023 Jan 1;52(1):e7-e20. doi: 10.1097/MPA.0000000000002215. PMID 37378896